CLINICAL TRIAL: NCT03129646
Title: An Open Label, Phase III, Randomized Controlled, Multicentre Non-Inferiority Trial to Compare Efficacy and Safety of Miltefosine and Paromomycin With SSG and PM Combination for Treatment of Primary Visceral Leishmaniasis (VL) Patients in Eastern Africa
Brief Title: Miltefosine/Paromomycin Phase III Trial for Treatment of Primary Visceral Leishmaniasis (VL) Patients in Eastern Africa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: The Netherlands Cancer Institute (Other); The Institute of Endemic Diseases (IEND), University of Khartoum (Unknown); Kenya Medical Research Institute (Other); Makerere University (Other); University of Gondar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-MILT/PM-01-VL
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2020-07

CONDITIONS: Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — miltefosine; Paromomycin; Antimony Sodium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 - MF/PM 14d (Experimental): Paromomycin 20 mg/kg/d IM for 14 days combined with oral miltefosine allometric dosing for 14 days
  Interventions: Drug: Miltefosine; Drug: Paromomycin
- Arm 2 - MF 28d/PM 14d (Experimental): Paromomycin 20 mg/kg/d IM for 14 days combined with oral miltefosine allometric dosing for 28 days
  Interventions: Drug: Miltefosine; Drug: Paromomycin
- Arm 3 - SSG/PM 17d (Active Comparator): Sodium Stibogluconate 20 mg/kg/day IM/IV combined with Paromomycin 15 mg/kg/day IM for 17 days
  Interventions: Drug: Paromomycin; Drug: Sodium stibogluconate

INTERVENTIONS:
Drug: Miltefosine — Miltefosine 10mg and 50mg capsules
  Other Names: Impavido
  Arms: Arm 1 - MF/PM 14d; Arm 2 - MF 28d/PM 14d
Drug: Paromomycin — Paromomycin sulfate equiv to 750mg paromomycin / 2ml amp
  Other Names: Paromomycin sulfate
Drug: Sodium stibogluconate — Sodium stibogluconate 33% 30 ml inj.
  Other Names: SSG
  Arms: Arm 3 - SSG/PM 17d

SUMMARY:
This is an open label, Phase III, randomized, controlled, parallel arm multicentre non-inferiority clinical trial to compare the efficacy and safety of two combination regimens of Miltefosine and Paromomycin with the standard SSG-PM for the treatment of primary adult and children VL patients in Eastern Africa.

DETAILED DESCRIPTION:
The 2 treatment regimens to be tested are:

* Arm 1: Paromomycin 20 mg/kg/d IM for 14 days combined with oral miltefosine allometric dosing for 14 days
* Arm 2: Paromomycin 20 mg/kg/d IM for 14 days combined with oral miltefosine allometric dosing for 28 days (recruitment in this arm was discontinued under protocol v4.0 dated 22 Jul 2019)

The reference arm is the current standard treatment for VL:

• Arm 3: Sodium Stibogluconate 20 mg/kg/day IM/IV combined with Paromomycin 15 mg/kg/day IM for 17 days

The target population will be VL patients from 4 to 50 years old in order to cover both paediatric and adult population.

Patients will be hospitalized for 14 days of PM and MF treatment for both arm 1 and arm 2. MF treatment will start at the same time as PM treatment and for arm 2 it will continue on an out-patient basis until completion of the 28 days treatment.

SSG&PM combination therapy will be administered for 17 days according to routine VL treatment guidelines and patients will remain hospitalized for the entire duration of the treatment.

All patients will be asked to return to the hospital for a full assessment on day 28, and for followup visits on day 56 and at six months.

To respond to the objectives, study assessments will be carried out at screening and on days 1, 3, 7, 14, 21, 28, 56 (one-month post-treatment) and 210 (six-month post-treatment). These assessments will include clinical, parasitological, haematological, biochemistry, safety, pharmacokinetic and pharmacodynamics assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical signs and symptoms of VL and confirmatory parasitological microscopic diagnosis
* Patients aged 4 to < 50 years who are able to comply with the study protocol.
* Patients for whom written informed consent has been obtained (if aged 18 years and over) or signed by parents(s) or legal guardian for patients under 18 years of age. In the case of minors, assent from the children also needs to be obtained as per each country regulatory requirements

Exclusion Criteria:

* Patients who are relapse cases
* Patients with Para-Kala azar dermal leishmaniasis grade 3
* Patients who have received any anti-leishmanial drugs in the last 6 months
* Patients with severe malnutrition (for children aged <5 years: weight-for-height WHO reference curves by sex, z score <-3; for children patients 5-18 years: BMI-for-age WHO reference curves by sex, z score < -3; for adults >18 years: BMI < 16)*
* Patients with positive HIV diagnosis
* Patients with previous history of hypersensitivity reaction or known drug class allergy to any of the study treatments
* Patients with previous history of cardiac arrhythmia or with a clinically significant abnormal ECG
* Patients suffering from a concomitant severe infection such as TB, schistosomiasis or any other serious underlying disease (e.g. cardiac, renal, hepatic) or chronic condition which would preclude evaluation of the patient's response to study medication
* Pregnant or lactating women
* Female patients of child bearing age who do not accept to have a pregnancy test done at screening and/or who do not agree to use contraception from treatment period until 5 months after the end of treatment (see section 15.2)
* Patients with haemoglobin < 5g/dl
* Patients with signs of severe VL according to Investigator's judgement, requiring an indication for AmBisome therapy based on the clinical manifestations (such as jaundice, bleeding, edema) and clinically significant abnormalities in the following laboratory parameters: haemoglobin, WBC, platelets, liver enzymes (ALT and AST), total bilirubin and creatinine
* Patients with pre-existing hearing loss based on audiometry at baseline
* Patients who cannot comply with the planned scheduled visits and procedures of the study protocol

  * Note: for Ethiopia only: Patients with severe malnutrition (for patients 4-18 years: MUAC cut-off based on MUAC-for-height reference table; for patients > 18 years: MUAC < 170 mm)

Ages: 4 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 439 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Definitive Cure | 6 months follow-up (Day 210)
  Cure at 6 months follow up defined as absence of clinical signs and symptoms of VL at D210 and no requirement for rescue treatment during the trial (e.g. no relapse or initial treatment failure).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From Screening to day 210
  1. Frequency of SAEs and AEs requiring treatment discontinuation
  2. Frequency and severity of adverse events from the start of treatment through the last visit, at day 210.
Initial cure at day 28 | Initial cure: day 28; Probable cure: day 56
  Initial cure: cure at the end of treatment (Day 28), defined as recovery of clinical signs and symptoms; absence of parasites (microscopy) and no rescue treatment administered up to and including Day 28.
  Probable cure: absence of clinical signs and symptoms of VL at D56 and no prior requirement for rescue medication.
Pharmacokinetics of paromomycin and miltefosine | During treatment, at 1 month (day 56) and 6 months (day 210) follow-up
  Total and partial blood plasma exposure to paromomycin and miltefosine defined as the area under the concentration-time curve
Pharmacodynamics | From baseline until day 210, and at any suspicion of relapse during the trial.
  Blood parasite clearance over time (qualitative and quantitative), as measured by qPCR from blood samples
Compliance to miltefosine treatment in an outpatient setting | Day 15 to day 28 miltefosine treatment
  Compliance to MF treatment in an outpatient setting will be assessed through patients' hospital records history, drug accountability and PK measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Mbui, MD, Principal Investigator — Kenya Medical Research Institute; Joseph Olobo, MD, Prof, Principal Investigator — College of Health Sciences, Makerere University, Uganda; Ahmed M Musa, MD, Prof, Principal Investigator — Institute of Endemic Diseases, Sudan; Rezika Mohammed, MD, Principal Investigator — University Hospital of Gondar, Ethiopia
Locations (7):
- Ethiopia (2):
  - Abdurafi MSF Health Center, Ābderafī, Amhara
  - University Hospital of Gondar, Gonder
- Kacheliba Hospital, Kapenguria, West Pokot County, Kenya
- Sudan (3):
  - El Hassan Centre for Tropical Medicine, Doka, Al Qaḑārif
  - Tabarak Allah MSF Hospital, Gedaref, Al Qaḑārif
  - Um El Kher Hospital, Gedaref
- Amudat Hospital, Amudat, Karamoja, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Musa AM, Mbui J, Mohammed R, Olobo J, Ritmeijer K, Alcoba G, Muthoni Ouattara G, Egondi T, Nakanwagi P, Omollo T, Wasunna M, Verrest L, Dorlo TPC, Musa Younis B, Nour A, Taha Ahmed Elmukashfi E, Ismail Omer Haroun A, Khalil EAG, Njenga S, Fikre H, Mekonnen T, Mersha D, Sisay K, Sagaki P, Alvar J, Solomos A, Alves F. Paromomycin and Miltefosine Combination as an Alternative to Treat Patients With Visceral Leishmaniasis in Eastern Africa: A Randomized, Controlled, Multicountry Trial. Clin Infect Dis. 2023 Feb 8;76(3):e1177-e1185. doi: 10.1093/cid/ciac643. PMID 36164254

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03129646/Prot_SAP_ICF_000.pdf